CLINICAL TRIAL: NCT05578352
Title: The Exploreration of the Management for the Positive IAA in Patients With Type 2 Diabetes After Premix Insulin Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-8-5-01
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral hyppoglycemia drug group (Active Comparator): Oral hyppoglycemia drugs, including metforemin, acarbose, dipeptidyl peptidase 4 inhibitors, or SGLT2-ihibitors, are added to reduce insulin dose.
  Interventions: Other: Add oral hyppoglycemia drug
- GLP-1RA group (Active Comparator): Add GLP-1 receptor agonists to reduce insulin dose.
  Interventions: Other: Add GLP-1 receptor agonist
- long-acting insulin group (Active Comparator): Change premix insulin to long-acting insulin plus oral hyppoglycemia drugs
  Interventions: Other: Change insulin
- Control group (No Intervention): continue the present premix insulin treatment, adjust insulin dose according to the bloog glucose profile in FGM to improve glycemic control.

INTERVENTIONS:
Other: Add oral hyppoglycemia drug — Oral hypoglycemic drugs with insulin sensitization effect are added, reduce insulin dose according to blood glucose
  Arms: Oral hyppoglycemia drug group
Other: Add GLP-1 receptor agonist — Add GLP-1 receptor agonist and reduce insulin dose according to blood glucose
  Arms: GLP-1RA group
Other: Change insulin — Change premix insulin to long-acting insulin
  Arms: long-acting insulin group

SUMMARY:
Premix insulin is widely used, with high proportion of positive insulin autoimmune antibody in patients with type 2 diabetes. The positive insulin autoimmune antibody may affect blood glucose control. We aim to explore the management for the positive insulin autoimmune antibody and blood glucose control in these patients, and investigate the immune cells changes with the change of different glucose lowering drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes;
* Treated with premix insulin, two or three injections a day, single drug or combination of oral hypoglycemic drugs;
* The treatment regimen was stable for more than 2 months;
* With positive insulin antibody

Exclusion Criteria:

* Patients treated with GLP-1 agonist in the last 3 months;
* Allergic to insulin;
* Impaired liver and renal function (ALT 2.5 times higher than the upper limit of normal value; serum creatinine was 1.3 times higher than the upper limit of normal);
* A history of drug abuse and alcohol dependence;
* Used systemic glucocorticoids therapy in recent 3 months;
* Patients with infection or stress within four weeks;
* Patients who cannot tolerate FGM;
* Pregnant or preparing to become pregnant;
* Considered unsuitable to participate by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Insulin autoimmune antibody | 3 month
  The change of insulin autoimmune antibody

SECONDARY OUTCOMES:
HbA1c | 3 month
  The change of glycated hemoglobin
Time in range | 3 month
  The change of time in range
Time below range | 3 month
  The change of time below range
B cell | 3 month
  the change of B cell subsets
T cell | 3 month
  the change of T cell subsets

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, Professor, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing Medical Univesity, Nanjing, China